CLINICAL TRIAL: NCT00663455
Title: A Multicenter, Randomized, Parallel-group, Trial to Reduce Toxicity of Calcineurininhibitor-therapy in Steroid-free Longterm Immunosuppression in Pediatric and Adolescent Kidney Transplant Recipients
Brief Title: Randomized Study to Reduce Calcineurininhibitor Toxicity in Pediatric and Adolescent Kidney Transplant Recipients
Acronym: Recaltox
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment goals were not achieved. Extension of the trial concept had to be abjected due to methodological reasons.
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Recaltox-1
Record Dates: First submitted 2008-04-21; First posted 2008-04-22 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Kidney Transplant
Keywords: kidney transplant recipients; children and adolescents with kidney transplants

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Other): Reduction of CSA-dosing over 4 months. Therapy control by safety parameters (serum creatinine, C2-monitoring, renal biopsy).
  Interventions: Drug: Reduction of cyclosporine A (CSA)-dosing
- B (No Intervention): Standard CSA-dosing without reduction. Therapy control by C2-monitoring.

INTERVENTIONS:
Drug: Reduction of cyclosporine A (CSA)-dosing — Reduction of CSA-dosing over 4 months. Therapy control by safety parameters (serum creatinine, C2-monitoring, renal biopsy).
  Arms: A

SUMMARY:
The purpose of this study is to determine if a safe reduction of cyclosporine A in pediatric and adolescent patients with stable renal graft function, reduces signs of calcineurin-inhibitor toxicity.

DETAILED DESCRIPTION:
Chronic transplant nephropathy is one of the major causes of graft loss after renal transplantation. Toxicity of calcineurin-inhibitors is suspected to be one cause for loss of graft function. Therefore reduction of cyclosporine A dosing can result in longer graft survival and better graft function in patients after renal-transplantation. However, reduction of immunosuppression can result in acute rejection episodes, although it is less likely in patients with stable graft function 12 months or longer after successful renal transplantation.

Therefore the aim of this randomized, controlled study in pediatric and adolescent renal transplant recipients, is to compare the impact of reduced cyclosporine A-dosing to standard CSA-dosing on renal graft function. Therapy monitoring in both groups will be performed by obtaining CSA blood levels two hours after intake, as they provide an individual insight in pharmacokinetics in comparison to conventional trough level (C0)-measurements.

Secondary objectives to evaluate are

1. the evaluation of the health-related Quality of life and psychosocial burden in the two treatment arms.
2. measurement of the NFAT-regulated gene expression (nuclear factor of activated t-cells) of intracellular cytokines [Interleukin-2, TNF-alpha, Interferon-gamma and GMCSF) by quantitative PCR as measurement of CSA activity.
3. To obtain new insights by screening for metabolites conjunct with clinic features of nephrotoxicity or graft rejections a metabolomic screening and a targeted analysis (trimethylamine-N-oxide, neopterin and kynurenine/tryptophan ratio) will be performed.

ELIGIBILITY:
Inclusion Criteria:

* age at inclusion 3-16 years
* male or female patients
* recipient of first or second renal transplant
* graft age > 24 months
* last acute rejection episode > 6 months ago
* Immune suppression comedication Mycophenolatmofetil (MMF) in a dose range of 1200 +/- 200 mg/m² BSA/d within at least 6 months or minimal MPA-AUC ≥ 45 mg x h/l. If MPA-AUC < 45 mg x h/l adjustment of dosage with re-screening in ≥ 4 weeks is possible.
* Application of CSA in stable dosing within the last 3 months before study inclusion and CSA-C2-level > 500 ng/ml. If CSA-C2-level < 500 ng/ml adjustment of dosage with re-screening in ≥ 4 weeks is possible.
* steroid-free immunosuppression for at least 6 months before enrollment
* biopsy of the renal graft without any signs of acute rejection (def. according to BANFF classification), within 3 months before enrollment
* written informed consent of parents/legal guardians and, if applicable, patient's consent

Exclusion Criteria:

* glomerular filtration rate < 40 ml/min/1.73 m2 BSA (acc. to Schwartz' formula) at time of enrollment
* > 2 episodes of acute graft rejection within 12 months prior to enrollment
* condition after steroid-resistant graft rejection
* actual participation in another clinical trial
* Recurrence of primary renal disease in the graft
* proven infection with EBV and/ or CMV and antiviral therapy within 3 months prior to enrollment
* proven infection with polyoma virus within 3 months prior to enrolment
* pregnant or nursing women
* hemoglobin < 8 g/dl at screening visit
* non-treated arterial hypertension
* uncontrolled infectious disease
* history of malignancy of any organ system, treated or non-treated

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2008-12; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Mean decline per month in glomerular filtration rate (calculated acc. to Schwartz' formula) during the clinical trial - comparison between the two study arms (CSA-dose reduction group and group with constant CSA-dosing) | 24 months

SECONDARY OUTCOMES:
Evaluation of the NFAT-regulated gene expression (nuclear factor of activated t-cells) of intracellular cytokines [Interleukin-2, TNF-alpha, Interferon-gamma and GMCSF) by quantitative PCR as measurement of CSA activity | 24 months
Health-related Quality of life evaluation using validated questionnaires (TACQoL) to determine differences between the two study arms | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jörg Dötsch, MD, Principal Investigator — Dept. of Pediatric Nephrology, University Hospital Erlangen, Germany
Locations (10):
- Germany (10):
  - Dept. of Pediatric Nephrology, University Hospital Erlangen, Erlangen
  - Dept. of Pediatric Nephrology, University Hospital Freiburg, Freiburg im Breisgau
  - Dept. of Pediatric Nephrology, University Hospital Hamburg, Hamburg
  - Dept. of Pediatric Nephrology, University Hospital Hannover, Hanover
  - Dept. of Pediatric Nephrology, University Hospital Heidelberg, Heidelberg
  - Dept. of Pediatric Nephrology, University Hospital Jena, Jena
  - Dept. of Pediatric Nephrology, Community Hospital Memmingen, Memmingen
  - Dept. of Pediatric Nephrology, University Hospital München, Munich
  - Dept. of Pediatric Nephrology, University Hospital Muenster, Münster
  - Dept. of Pediatric Nephrology, University Hospital Rostock, Rostock